CLINICAL TRIAL: NCT05294224
Title: The Relationship Between Disease Severity and Various Lower Extremity Parameters in Individuals With Knee Osteoarthritis
Status: Completed | Type: Observational
Sponsor: Dilara Özen Oruk (Other)
Collaborators: Muğla Sıtkı Koçman University (Other)
Responsible Party: Sponsor-Investigator, Dilara Özen Oruk, Research Assistant, Muğla Sıtkı Koçman University
Organization: Muğla Sıtkı Koçman University (Other)
Other Study IDs: 210077/10
Record Dates: First submitted 2022-03-15; First posted 2022-03-24 (Actual); Last update posted 2024-03-15 (Actual); Status verified 2024-03

CONDITIONS: Knee Osteoarthritis; Knee Injuries
Keywords: muscle thikness; cartilage thickness; balance; postural stability; kinesiophobia; gait; degeneration; function
MeSH Terms: conditions — Osteoarthritis, Knee; Knee Injuries; Kinesiophobia

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study perform to investigate the relationship between quadriceps femoris (QF) strength, QF thickness, femoral cartilage thickness, knee function, balance, kinesiophobia and gait of the patients with knee osteoarthritis.

DETAILED DESCRIPTION:
Osteoarthritis (OA) is one of the most common chronic degenerative diseases in the world, which progresses slowly, can cause pain, stiffness and dysfunction, and reduces the quality of life.

OA is particularly common in weight-bearing joints such as the knee and the functional status of patients with OA is adversely affected various factors such as immobility due to pain, decrease in muscle strength and joint range of motion, etc.

In relation to this, walking difficulty and decrease in walking speed, balance problems and an increase in the risk of falling are a picture that can be encountered in the later stages of the disease.

The aim of this study is to investigate the relationship between QF strength, QF thickness, femoral cartilage thickness, knee function, balance, kinesiophobia and gait of the patients with knee OA.

ELIGIBILITY:
Inclusion Criteria:

* Volunteer patients who applied to the Physical therapy and Rehabilitation department with knee pain

Exclusion Criteria:

* Individuals who have received intra-articular therapy for gonarthrosis in the last 6 months, who have undergone arthroscopic surgery, and who have additional pathologies in their lower extremities
* Individuals with physical, mental and/or psychological disorders that may affect participation in the study

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Volunteer patients who applied to the Physical therapy and Rehabilitation department with knee pain
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2022-04-17 (Actual); Primary Completion 2022-08-30 (Actual); Study Completion 2023-09-30 (Actual)

PRIMARY OUTCOMES:
QF muscle thickness | Day 1
  QF muscle thickness
QF muscle strength | Day 1
  QF muscle strength
Femoral cartilage thickness | Day 1
  Femoral cartilage thickness
Knee function | Day 1
  Knee function assessment with The Knee injury and Osteoarthritis Outcome Score (KOOS). It is a 42-item questionnaire, including 5 subscales: symptoms, pain, ADLs, sports/recreation, and quality of life. The maximum score a patient can achieve is 100, indicating no knee problems. The minimum score is zero, indicating severe knee problems.
Kellgreen-Lawrence Radiological Stages | Day 1
  Kellgreen-Lawrence Radiological Stages:
  Grade 1 (doubtful): doubtful joint space narrowing and possible osteophytic lipping. grade 2 (minimal): definite osteophytes and possible joint space narrowing. grade 3 (moderate): moderate multiple osteophytes, definite narrowing of joint space and some sclerosis and possible deformity of bone ends.
Kinesiophobia | Day 1
  Tampa Kinesiophobia Scale: The total score of the scale range from 17- 68, where 17 means no kinesiophobia, 68 means severe kinesiophobia, and score ± 37 indicates there is kinesiophobia.
Balance and gait | Day 1
  Tinetti Score: It uses a 3-point ordinal scale of 0, 1 and 2. Gait is scored over 12 and balance is scored over 16 totalling 28. The lower the score on the Tinetti test, the higher the risk of falling.
Low Extremity Functionality and Fall Risk | Day 1
  30 sec sit to stand test

CONTACTS AND LOCATIONS:
Locations (1):
- Mugla Sıtkı Koçman University, Muğla, Turkey (Türkiye)